CLINICAL TRIAL: NCT00691652
Title: Phase I/II Study of Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Brief Title: Clofarabine and Rituximab in Treating Patients With Relapsed Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding ended when only one subject enrolled and subject withdrew early.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000597410; P30CA069533 (NIH); OHSU-HEM-07156-L; IRB#4101; GENZYME-OHSU-HEM-07156-L
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma
Keywords: extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; cutaneous B-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Clofarabine; DNA Methylation; Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction; Chromatography, High Pressure Liquid

ARMS (1):
- Oral Clofarabine + Rituximab in Relapsed B Cell NHL (Experimental): Phase I: Oral Clofarabine x 14 days for up to 8 cycles at assigned dose level below (1 cycle equals 14 days on drug, 14 days off).
  Rituximab weekly for 4 weeks than monthly for up to 8 cycles on day 1 of cycle 375 mg/m2 IV
  Dose Level 1: 2 mg Dose Level 2: 4 mg Dose Level 3: 6 mg
  Phase II:
  Oral Clofarabine x 14 days for up to 8 cycles (Dose determined from phase I) AND Rituximab weekly for 4 weeks than monthly for up to 8 cycles on day 1 of cycle 375 mg/m2 IV
  Interventions: Biological: rituximab; Drug: clofarabine; Genetic: DNA methylation analysis; Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: polymerase chain reaction; Other: high performance liquid chromatography; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Administered weekly times 4 weeks and then monthly during the study for up to 8 cycles and will be given on day 1 of clofarabine. A peripheral or central intravenous (IV) line will be established. The initial dose rate at the time of the first infusion should be 50/mg/hr for the first hour. If no toxicity is seen, the dose rate may be gradually escalated (50 mg/hr increments at 30 minute intervals) to a maximum of 300 mg/hr. If the first dose of rituximab is well tolerated, the starting flow rate for the administration of subsequent doses will be 100 mg/hr then gradually increased (100 mg/hr increments at 30 minute intervals) not to exceed 400 mg/hr.
Drug: clofarabine — Phase 1 dosing: Initially, 3 patients will be enrolled into a dose level during the dose escalation portion. Level 1: 2mg fixed dose times 14 days for up to 8 cycles. Level 2: 4mg fixed dose times 14 days for up to 8 cycles. Level 3: 6mg fixed dose times 14 days for up to 8 cycles. Phase II dosing: The phase II dose of oral clofarabine will be determined from the phase 1.
Genetic: DNA methylation analysis — We will use an HPLC assay developed by Yu et al31 to determine the DNA methylation (DMI) index in peripheral blood and bone marrow of patients entering this trial and after treatment with clofarabine and rituxan
Genetic: gene expression analysis — Total RNA will be processed for determination of gene expression by microarray
Genetic: microarray analysis — we will scan the microarray slides with an Axon scanner, and quantify data using the GeneSight software. Local background is subtracted and data points with no signal, high background, or spot asymmetry are eliminated. We will adjust genes with low expression and low signal intensity to a minimal raw value of 5: This avoids unwarranted mathematical distortions due to division by decimals << 1. After calculating the ratio of the Cy5 /Cy3 fluorescence signal intensity for each gene, we normalize the data relative to the mean intensity from all genes.
Genetic: polymerase chain reaction
Other: high performance liquid chromatography — Fifteen µg of DNA will be sonicated for 60 seconds on ice into 200 bp-1000 bp fragments. Samples are then denatured at 1000C for 5 minutes and cooled on ice to prevent re-annealing. Sixty units of nuclease S1 (Invitrogen) and 112.5 mu of snake venom phosphodiesterase I (Sigma) in 12 µl of S1 dilution buffer is then added to the samples and incubated at 370C for 18 hours. Samples are reheated to 1000C for 5 minutes, snap cooled again on ice, and another sixty units of nuclease S1 and 112.5 mu of snake venom phosphodiesterase I are added and incubated at 370C for another 4 to 6 hours. The pH of each sample was raised to 8.5 with 0.5 M Tris, pH 10. Two and a half units of alkaline phosphatase (Sigma) are added and incubated for 2 additional hours at 370C. One hundred µl of 0.05M potassium phosphate, pH 7 is added to final samples before 50 µl of the clear supernatant is injected into the reverse-phase high performance liquid chromatography (HPLC).
Other: laboratory biomarker analysis — 50 µl of the clear supernatant is injected into the reverse-phase high performance liquid chromatography (HPLC).
  Other Names: High Performance Liquid Chromatography (HPLC)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving clofarabine together with rituximab may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of clofarabine when given together with rituximab and to see how well they work in treating patients with relapsed B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of clofarabine in adult patients with relapsed CD20-positive B-cell non-Hodgkin lymphoma (NHL).
* To estimate objective response rates of clofarabine in combination with rituximab in these patients.

Secondary

* To determine the 1-year progression-free survival of this regimen using the mean tolerated dose in these patients.
* To determine the safety and efficacy of this regimen in these patients.
* To determine if clofarabine acts as an inhibitor of DNA methylation similar to cladribine by performing scientific correlates.
* To determine whether response to clofarabine alone or in combination with rituximab correlates with changes in global serum DNA methylation index.
* To identify the gene activated by clofarabine therapy by using genomic DNA and RNA array technology.

OUTLINE: This is a phase I, dose-escalation study of clofarabine followed by a phase II study.

Patients receive oral clofarabine once daily on days 1-14 of all courses and rituximab IV on days 1, 8, 15, and 22 of course one and then on day 1 of courses 2-8. Courses repeat every 4 weeks. After 2 courses of therapy, patients who are eligible for stem cell transplantation may either undergo transplantation or continue receiving study drugs until disease progression or unacceptable toxicity for up to a total of 8 courses of treatment.

Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed to identify global DNA methylation differences and correlate changes in methylation index (MI) with patient outcome after treatment with clofarabine with or without rituximab via high performance liquid chromatography (HPLC); to determine differences in gene expression via microarray analysis and micro-RNA (miRNA) expression via quantitative polymerase chain reaction (PCR) in patients with high compared to low global DNA methylation index and miRNA expression for CD5+ B-lymphocytes obtained from pediatric tonsils and from B-lymphocytes of 5 healthy controls; and to determine gene expression and miRNA profiles in patients before and after treatment with clofarabine with or without rituximab via genomic DNA arrays.

After completion of study treatment, patients are followed once a year for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed B-cell lymphoma

  * Relapsed disease
  * CD20-positive disease
* Must have had bone marrow aspiration and biopsy (uni- or bilateral) within the past 42 days and chest CT and CT of the abdomen and pelvis within the past 28 days
* Documented bidimensionally measurable disease within the past 28 days

  * Patients with non-measurable disease in addition to measurable disease must have all non-measurable disease assessed within 42 days prior to registration

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group(ECOG) performance status 0-2
* Leukocyte count ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after completion of study therapy
* No known AIDS or HIV-associated complex
* No active hepatitis B infection
* No other severe concurrent disease, history of serious organ dysfunction, or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* No uncontrolled systemic fungal, bacterial, viral, or other infection, defined as ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment
* No history of intolerance or allergic reactions to clofarabine or rituximab
* No significant concurrent disease, illness, or psychiatric disorder that would compromise the patient's safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* No concurrent active GI disease that may impair absorption of oral clofarabine

PRIOR CONCURRENT THERAPY:

* Recovered from all previous therapies
* No prior gastrointestinal (GI) surgery that may impair absorption of oral clofarabine
* More than 2 weeks since prior and no concurrent anticancer therapy, except for hydroxyurea
* More than 4 weeks since prior radioimmunotherapy
* More than 1 month since prior investigational agents
* No concurrent cytotoxic therapy or investigational therapy
* No other concurrent investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy
* No concurrent alternative medications (e.g., herbal or botanical for anticancer purposes)
* No other concurrent chemotherapy or immunotherapy
* No concurrent radiotherapy
* No concurrent colony stimulating factors (phase I portion of the study)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Okada, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (4.949)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of Oral Clofarabine in Adult Patients With Relapsed CD20+ Non-Hodgkin Lymphoma(NHL)
Description: Initially, 3 patients will be enrolled into a dose level during the dose-escalation portion:
  * If no patient experiences dose-limiting toxicities during the first 4 weeks, then 3 patients will be enrolled into the next dose level.
  * If one of the three patients develops dose-limiting toxicities, then 3 additional patients will be enrolled in that cohort. If none of the additional 3 patients experiences dose-limiting toxicities, then further dose-escalation occurs.
  * If one additional patient experiences dose-limiting toxicities, then the maximum tolerated dose is exceeded.
Time Frame: 14 days for up to 8 cycles (1 cycle equals 14 days on drug, 14 days off drug) for a total of up to 224 days
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

2. Primary Outcome: Estimate Objective Response Rates of Oral Clofarabine in Combination With Rituximab in Relapsed CD20+NHL
Time Frame: Oral Clofarabine x 14 days for up to 8 cycles (1 cycle equals 14 days on drug, 14 days off drug) for a total of up to 224 days AND Rituximab weekly for 4 weeks than monthly for up to 8 cycles on day 1 of cycle
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine One-year Progression Free Survival Using the MTD of Clofarabine With Rituximab in Relapsed CD20+NHL
Time Frame: One year after study drug(s) have been given. Duration of study up to 1 year.
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

4. Secondary Outcome: Determine the Safety and Efficacy of Clofarabine in Combination With Rituximab
Time Frame: Duration of the study, up to 1 year.
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

5. Secondary Outcome: Whether Clofarabine Acts as an Inhibitor of DNA Methylation Similar to Cladribine by Performing Scientific Correlates
Time Frame: Duration of the study, up to 1 year.
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

6. Secondary Outcome: Whether Response to Clofarabine Alone or in Combination With Rituximab Correlates With Changes in Global Serum DNA Methylation Index
Time Frame: Duration of the study, up to 1 year.
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

7. Secondary Outcome: Identity of the Gene Activated by Clofarabine Therapy by Using Genomic DNA and RNA Array Technology
Time Frame: Twice monthly at standard of care visits for 3 months post last cycle of chemotherapy.
Population: Insufficient data to analyze outcome. Funding ended when only one subject enrolled and subject withdrew early.
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Oral Clofarabine + Rituximab in Relapsed B Cell NHL
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No